CLINICAL TRIAL: NCT02411214
Title: Fertility Preservation in the Male Pediatric Population: a Patient and Parent Perspective of Factors Influencing the Decisional Process
Brief Title: Decisional Process in Male Fertility Preservation
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Wyns, Head of department gynecology-andrology, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: FP1
Record Dates: First submitted 2015-04-02; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Infertility; Quality of Life; Cancer
MeSH Terms: conditions — Infertility; Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- <12 years: children under 12 years diagnosed with cancer questionnaire survey
  Interventions: Other: survey
- 12-18 years: adolescents diagnosed with cancer questionnaire survey
  Interventions: Other: survey
- parents: parents of children and adolescents diagnosed with cancer questionnaire survey
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — questionnaire survey sent by regular mail for 3 groups

SUMMARY:
The survey analyses how to improve the decision-making process for fertility preservation in the pediatric population based on

1. patient and parent feelings about fertility preservation counselling
2. influence of the emotional state of patients and parents on fertility preservation acceptance
3. support of medical staff and family The study revealed that attention to the fertility preservation pathways was important for the satisfaction of patient's and parent's expectations

DETAILED DESCRIPTION:
Questionnaire survey via regular mail to an eligible population (boys and adolescents aged 0 to 18 years diagnosed with cancer at the Cliniques universitaires Saint Luc) between January 2005 and May 2013.

Three different questionnaires, for children (<12 years and 12-18 years) and parents respectively, established based on information from focus groups and subsequently reviewed by the institutional ethics board before being sent.

ELIGIBILITY:
Inclusion Criteria:

* prepubertal boys and adolescents diagnosed with cancer in a university hospital setting between january 2005 and may 2013

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: prepubertal boys and adolescents diagnosed with cancer in a university hospital setting between january 2005 and may 2013 and their parents
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
factors improving the decision-making process for fertility preservation | less than 1 year
  factors improving the decision-making process for fertility preservation assessed by three specific questionnaires (parent, adolescent and children)

SECONDARY OUTCOMES:
patient and parent feelings about fertility counseling | less than 1 year
  patient and parent feelings about fertility counseling assessed by three specific questionnaires (parent, adolescent and children)
influence of the emotional state of parents and patients on fertility preservation acceptance | less than 1 year
  influence of the emotional state of parents and patients on fertility preservation acceptance assessed by three specific questionnaires (parent, adolescent and children)
support of medical staff and family | less than 1 year
  support of medical staff and family assessed by three specific questionnaires support of medical staff and family (parent, adolescent and children)

REFERENCES:
- [Derived] Wyns C, Collienne C, Shenfield F, Robert A, Laurent P, Roegiers L, Brichard B. Fertility preservation in the male pediatric population: factors influencing the decision of parents and children. Hum Reprod. 2015 Sep;30(9):2022-30. doi: 10.1093/humrep/dev161. Epub 2015 Jul 3. PMID 26141713